CLINICAL TRIAL: NCT01155544
Title: Improving Outcomes in Psychosis Associated With Substance Use Using Aripiprazole
Acronym: SIP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Seems to have simply stopped.
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-160B
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Substance Abuse; Substance Dependence
Keywords: Aripiprazole; Psychotic experiences; Substance abuse; Substance dependence; Craving; Mood; Substance use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole (Active Comparator)
  Interventions: Behavioral: Behavioral Intervention
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Behavioral Intervention

INTERVENTIONS:
Behavioral: Behavioral Intervention — Preventing recurrence of substance use.

SUMMARY:
This project focuses on the under-researched group of individuals who develop psychotic episodes of short duration (less than four weeks) while using substances. This includes individuals diagnosed with psychotic disorder not otherwise specified (PNOS) or substance-induced psychotic disorder (SIP) AND substance abuse or dependence. Very little is known about the most appropriate maintenance/relapse prevention management of these subjects. These individuals are not diagnosed with a primary psychosis because psychotic symptoms are too short-lived or non-specific, the onset of substance use precedes the onset of psychotic symptoms and the subject has not experienced sufficient psychotic symptoms in the absence of substance use. However, previous studies have shown that they are at high risk of recurrence of psychotic symptoms. Thus, this project will assess the efficacy of the second-generation antipsychotic aripiprazole for maintenance treatment of subjects who had a recent psychotic episode of short duration associated with substance use. The investigators will compare aripiprazole and placebo for preventing the recurrence of psychotic symptoms and decreasing substance use during a 6-month maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-defined diagnosis of psychosis NOS or substance-induced psychosis assessed with the Structured Clinical Interview for Axis I DSM-IV Disorders (SCID-I/P) (First 1998)
* onset of psychotic symptoms following onset of substance use
* current DSM-IV-defined diagnosis of substance abuse or dependence assessed with the SCID-I/P
* duration of the acute psychotic episode less than 4 weeks
* aged 16 to 44
* competent and willing to sign informed consent
* for women, a negative urine pregnancy test and agreement to use a medically accepted method of birth control and not to become pregnant during the study
* at the entry of the maintenance phase, remission of psychotic symptoms defined as 1) simultaneous ratings of <3 ("mild) on all of the following Brief Psy¬chiatric Rating Scale-Anchored version items (BPRS-A; Woerner et al. 1988): suspiciousness, unusual thought content, hallucinations, conceptual disorganization; and 2) a Clinical Global Impressions Scale (CGI; Guy 1976) Se-verity rating of 3 ("mild") or less.

Exclusion Criteria:

* DSM-IV criteria for schizophrenia, schizophreniform disorder, schizoaffective disorder, a psychotic disorder due to a general medical condition, shared psychotic disorder, or a major mood disorder (major depression or bipolar mania) with psychotic features
* antipsychotic treatment for more than six months prior to enrollment
* serious neurological or endocrine disorder or any medical condition or treatment known to affect the brain
* medical condition that requires treatment with a medication that has psychotropic effects
* significant risk of suicidal or homicidal ideation or behavior
* cognitive or language limitations, or any other factor that would preclude subjects providing informed consent or participating in study procedures
* history of treatment resistance to aripiprazole
* medical contraindications to aripiprazole
* hypersensitivity to aripiprazole or any component of the products.

Ages: 16 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Psychotic Symptoms | 7 months
  Psychotic symptoms wil be assessed with the Structured Interview for Prodromal Symptoms and the Brief Psychiatric Rating Scale. We will focus on time to first recurrence of psychotic symptoms and rate of recurrence.
Frequency/amount of substance use | 7 months
  Frequency and amount of cannabis and other substance use will be recorded with the Timeline Follow-Back Method. We will focus on time to first recurrence of substance use and rate of recurrence.

SECONDARY OUTCOMES:
Mood symptoms | 7 months
  Mood symptoms will be assessed with the Hamilton Depression Rating Scale
Adverse Events | 7 months
  Adverse events will be assessed with the Systematic Assessment for Treatment Emergent Events interview, Simpson-Angus Scale for Extrapyramidal Symptoms, the Abnormal Involuntary Movement Scale, the Barnes Akathisia Scale, and blood tests (fasting glucose, insulin and lipid profile tests)

CONTACTS AND LOCATIONS:
Overall Officials: Serge Sevy, MD, MBA, Principal Investigator — Feinstein Institute for Medical Research
Locations (2):
- United States (2):
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - North Shore Hospital, Manhasset, New York